CLINICAL TRIAL: NCT01264679
Title: An Open-Label Extension Study of the Safety and Efficacy of Ferumoxytol for the Episodic Treatment of Iron Deficiency Anemia in Pediatric Subjects With Chronic Kidney Disease
Brief Title: A Trial of Ferumoxytol for the Episodic Treatment of Iron Deficiency Anemia in Pediatric Participants With Chronic Kidney Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Several factors contributed to significant challenges in enrollment and led the Sponsor to discontinue the AMAG-FER-CKD-253 study as designed.
Sponsor: AMAG Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMAG-FER-CKD-253
Record Dates: First submitted 2010-12-20; First posted 2010-12-22 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-03

CONDITIONS: Iron Deficiency Anemia
Keywords: Iron deficiency anemia; Feraheme; ferumoxytol; chronic kidney disease; CKD; pediatric; dialysis-dependent; nondialysis-dependent
MeSH Terms: conditions — Anemia, Iron-Deficiency; Renal Insufficiency, Chronic | interventions — Ferrosoferric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ferumoxytol (Experimental): When a participant has persistent or recurrent IDA (defined as hemoglobin <12.0 grams [g]/deciliter [dL] and with either transferrin saturation <40% or ferritin <100 nanograms/milliliter), the participant will begin a 7-week treatment period. Participants will receive 2 IV injections of ferumoxytol 7.0 milligrams (mg) iron/kilogram (maximum of 510 mg/dose), the first dose administered on Day 1 and the second on Days 3 through 9 of the Treatment Period.
  Interventions: Drug: Ferumoxytol

INTERVENTIONS:
Drug: Ferumoxytol — IV Ferumoxytol
  Other Names: Feraheme

SUMMARY:
Study AMAG-FER-CKD-253 is an extension study of the combined AMAG-FER-CKD-251 (NCT01155375) and AMAG-FER-CKD-252 (NCT01155388) studies to evaluate the efficacy and safety of episodic treatment of iron deficiency anemia (IDA) with ferumoxytol.

DETAILED DESCRIPTION:
Study AMAG-FER-CKD-251 was a study evaluating the efficacy and safety of intravenous (IV) ferumoxytol in pediatric participants with dialysis-dependent chronic kidney disease (CKD). Study AMAG-FER-CKD-252 was a study evaluating the efficacy and safety of IV ferumoxytol in pediatric participants with nondialysis-dependent chronic kidney disease.

Due to significant challenges with enrollment for both studies, Study AMAG-FER-CKD-252 was combined with Study AMAG-FER-CKD-251 and enrollment continued under Study AMAG-FER-CKD-251.

Participants were enrolled by age cohorts in a stepwise manner following a safety review by the Data Safety Monitoring Board of 1 age cohort prior to enrollment of a subsequent age cohort, with progression from oldest to youngest: Randomization was stratified by the following age cohorts: 12 to <18 years, 6 to <12 years, 2 to <6 years, and 6 months to <2 years.

Participants who completed the combined AMAG-FER-CKD-251 and AMAG-FER-CKD-252 studies had the option of participating in this extension study.

ELIGIBILITY:
Key Inclusion Criteria include:

1. Participants who had completed participation in the combined AMAG-FER-CKD-251 and AMAG-FER-CKD-252 studies within 4 weeks of screening
2. Female participants of childbearing potential who are sexually active must be on an effective method of birth control and agree to remain on birth control until completion of participation in the study
3. Participant and/or legal guardian is capable of understanding and complying with the protocol requirements and is available for the duration of the study

Key Exclusion Criteria include:

1. Experienced a serious adverse event related to IV iron therapy in the combined AMAG-FER-CKD-251 and AMAG-FER- CKD-252 studies
2. Hemoglobin level ≤7 g/dL

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2011-12-27 (Actual); Primary Completion 2015-04-24 (Actual); Study Completion 2015-04-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- AMAG Pharmaceuticals, Inc., Waltham, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ferumoxytol: When a participant had persistent or recurrent iron deficiency anemia (IDA) (defined as hemoglobin <12.0 grams [g]/deciliter [dL] and with either transferrin saturation [TSAT] <40% or ferritin <100 nanograms [ng]/milliliter [mL]), the participant began a 7-week treatment period. Participants received 2 intravenous (IV) injections of ferumoxytol 7.0 milligrams [mg] iron (Fe)/kilogram (kg) (maximum of 510 mg/dose), the first dose administered on Day 1 and the second on Days 3 through 9 of the Treatment Period.
Period: Overall Study
Arm/Group | Ferumoxytol
Started | 8
Received at Least 1 Dose of Study Drug (Participants included in Safety and Intent-to-Treat (ITT) populations.) | 7
Completed | 3
Not Completed | 5
Not completed — Participation in Another Clinical Trial | 1
Not completed — Physician Decision | 1
Not completed — Sponsor's Suspension of Dosing | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: The Safety Population included all randomized participants who had received at least 1 dose of study drug.
Groups:
- Ferumoxytol: When a participant had persistent or recurrent IDA (defined as hemoglobin <12.0 g/dL and with either TSAT ≤40% or ferritin <100 ng/mL), the participant began a 7-week treatment period. Participants received 2 IV injections of ferumoxytol 7.0 mg Fe/kg (maximum of 510 mg/dose), the first dose administered on Day 1 and the second on Days 3 through 9 of the Treatment Period.
Arm/Group | Ferumoxytol
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The birth date is missing for 1 of the 7 pediatric participants. Therefore, mean and standard deviation for Age, Continuous is based on 6 participants.
  years
    number analyzed (Participants) | 6
    (all) | 15.3 (1.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 4
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change In Hemoglobin From Baseline To Week 5
Description: Mean changes in hemoglobin following the first course of ferumoxytol from Baseline to Week 5 were to be presented. Despite efforts to complete the studies as designed, several factors contributed to significant challenges in enrollment and led the Sponsor to discontinue the combined AMAG-FER-CKD-251 and AMAG-FER-CKD-252 studies, and the AMAG-FER-CKD-253 study. Blood samples were collected, but not run through an analysis to obtain outcome measure data. As such, the data set for this primary outcome measure cannot be summarized nor can the statistical analysis, as described in the protocol, be provided in a way that will provide any significant data based upon the limited study datasets.
Time Frame: Baseline, Week 5
Population: ITT Population included all randomized participants who had received at least 1 dose of study drug. Sample data were collected, but not run through any analysis to obtain outcome measure data. As such, summary of the data set is not possible.
Arm/Group | Ferumoxytol
Number analyzed (Participants) | 0

2. Secondary Outcome: Proportion Of Participants With An Increase In Hemoglobin From Baseline To Week 5 And To Week 7
Description: The proportion of participants with an increase hemoglobin to ≥1.0 g/dL or to ≥12.0 g/dL during the period from Baseline to Week 5 and to Week 7 following each course of ferumoxytol was to be presented. However, despite efforts to complete the studies as designed, several factors contributed to significant challenges in enrollment and led the Sponsor to discontinue the combined AMAG-FER-CKD-251 and AMAG-FER-CKD-252 studies, and the AMAG-FER-CKD-253 study. Blood samples were collected, but not run through an analysis to obtain outcome measure data. As such, the data set for this secondary outcome measure cannot be summarized in a way that will provide any significant data based upon the limited study datasets.
Time Frame: Baseline, Week 5 and Week 7
Population: as for outcome 1
Groups:
- Ferumoxytol: When a participant had persistent or recurrent IDA (defined as hemoglobin <12.0 g/dL and with either TSAT ≤40% or ferritin <100 ng/mL), the participant began a 7-week treatment period. Participants received 2 IV injections of ferumoxytol 7.0 mg Fe/kg (maximum of 510 mg/dose /dose), the first dose administered on Day 1 and the second on Days 3 through 9 of the Treatment Period.
Arm/Group | Ferumoxytol
Number analyzed (Participants) | 0

3. Secondary Outcome: Mean Change In TSAT From Baseline To Week 5 And To Week 7
Description: Mean changes in TSAT following the first course of ferumoxytol from Baseline to Week 5 and to Week 7 were to be presented. However, despite efforts to complete the studies as designed, several factors contributed to significant challenges in enrollment and led the Sponsor to discontinue the combined AMAG-FER-CKD-251 and AMAG-FER-CKD-252 studies, and the AMAG-FER-CKD-253 study. Blood samples were collected, but not run through an analysis to obtain outcome measure data. As such, the data set for this secondary outcome measure cannot be summarized in a way that will provide any significant data based upon the limited study datasets.
Time Frame: Baseline, Week 5 and Week 7
Population: as for outcome 1
Arm/Group | Ferumoxytol
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Randomization up to 24 months
Arm/Group | Ferumoxytol
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 3/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ferumoxytol (N=7)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Device breakage (General disorders) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ferumoxytol (N=7)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 (1)
Congestive cardiomyopathy (Cardiac disorders) | 1 (1)
Ventricular flutter (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Peritoneal lesion (Gastrointestinal disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (8)
Oral herpes (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1)
Procedural vomiting (Injury, poisoning and procedural complications) | 1 (1)
Ureteric anastomosis complication (Injury, poisoning and procedural complications) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (3)
Anuria (Renal and urinary disorders) | 2 (2)
Bladder spasm (Renal and urinary disorders) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1)
Air embolism (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
While sample data were collected, it was not run through any analysis to obtain the necessary outcome measure data. As such, summary of the data set is not possible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If there is no multi-site publication within 18 months after the Study has been completed or terminated at all Study sites, and all data has been received by Sponsor, the Site and SMO shall have the right to publish its results from the Study for non-commercial purposes, if submitted to Sponsor for review 60 days prior to submission of publication. Publication must remove all confidential information and may be delayed by up to 120 days to allow Sponsor to protect its interests.